CLINICAL TRIAL: NCT00695552
Title: DEMO II: A Randomized, Parallel-group, Observer-blinded Clinical Trial of Aerobic Exercise Versus Stretching Exercise for Patients With Light to Moderate Depression
Brief Title: The Effect of Exercise on Depressive Symptoms in Unmedicated Patients
Acronym: DEMOII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment process were slower than expected. Not enough money to continoue
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Merete Nordentoft, Professor, DMSc., Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEMOII
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Major Depression
Keywords: Major depression, exercise
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aerobic exercise on stationary bikes. Three sessions/week for 3 three months. First month the workload is equivalent to 65% of HRmax, the second month the workload is equivalent to 70% of HRmax, and the third month the workload is equivalent to 75% of HRmax
  Interventions: Behavioral: Aerobic exercise
- 2 (Placebo Comparator): Participants meets 3 times/week for 3 months. They will engage in low impact activities such as stretching exercises.
  Interventions: Behavioral: Low impact exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Aerobic exercise on stationary bikes. Three sessions/week for 3 three months. First month the workload is equivalent to 65% of HRmax, the second month the workload is equivalent to 70% of HRmax, and the third month the workload is equivalent to 75% of HRmax
  Arms: 1
Behavioral: Low impact exercise — Participants meets 3 times/week for 3 months. They will engage in low impact activities such as stretching exercises
  Arms: 2

SUMMARY:
This trial investigates the biological effect of exercise training on depression. Participants will randomly be allocated to either a aerobic exercise group performing exercise on stationary bikes or a group performing low-impact exercise such as stretching exercises. Both groups will attend sessions three times per week for 3 months. Before and after the intervention the investigators will measure the severity of depression using the Hamilton depression rating scale (HAM-D17).

DETAILED DESCRIPTION:
The yearly incidence of depression is estimated to be 3-5%, with a lifetime prevalence of 17% in western societies.Furthermore, Major depression is associated with increased mortality from somatic disorders such as cardiovascular disease, stroke, and endocrinological diseases. WHO and others stated that unipolar depressive disorders was the leading cause of disease burden in the western world in 2002 accounting for 9,0% of all disability adjusted life years. Projecting the current development in disease patterns unipolar depression is expected to be the second highest cause of global disease burden in 2030. With remission rates of approximately 50% using medical antidepressant therapy, the search for alternative or augmentation therapy is a key issue in depressive research.

In 2001 a meta-analysis concluded that the effect of exercise training could not be determined due to lack of good quality research. The authors found that the majority of trials were without blinded outcome assessment, lacked intention-to-treat analysis, and most had short follow-up. In this context, one of the authors in 2004 launched a pragmatic randomized controlled trial investigating the effect of exercise training on depressive symptoms - the DEMO trial(10). The 165 included participants were randomized to either aerobic, non-aerobic, or relaxation training in a four-month training programme. The primary outcome was the Hamilton depression rating scale (HAM-D17) and data collection ended June 1st 2007. After four month intervention there were no overall effect of exercise on depressive symptoms; the estimate at four month between non-aerobic and relaxation training was -0.9 (95%CI: -3.2 to 1.4) and between aerobic and relaxation training was 0.99 (95%CI: -1.3 to 3.3). These results do not support any biological effect of exercise on major depression. However, the majority (115/165) of patients had received antidepressant medication for more than six weeks at baseline thus the lack of a positive result could partly be explained by a treatment resistant group. A subgroup analysis of patients not medicated at baseline estimated the effect between non-aerobic and relaxation training to -1.7 (95% CI: -6.0 to 2.5) and between aerobic and relaxation training to 0.3 (95% CI: -3.9 to 4.6). The number of patients in this important sub-group, means that any conclusion on non-medicated patients is underpowered. In addition the literature suggest that the possible effect of exercise on depression is frequency and intensity related. In the DEMO trial the participants only trained twice pr. week.

This result from the DEMO trial is somewhat in contrast with the abundant publications of animal research showing that exercise stimulates hippocampal neurogenesis and in theory improves depressive symptoms and cognitive skills. The hippocampus is involved in cognitive functions such as memory and learning processes as well as regulation of the hypothalamus. In depression and neurodegenerative diseases such as Alzheimer and Parkinson Disease, which share features like impaired memory and learning abilities, the hippocampus is characterized by atrophia. In addition to a decreased hippocampal volume, brain imaging studies have observed reduction in volume of prefrontal cortex of depressed patients, though postmortem studies have less evident results.

Prospective studies on healthy adults suggest that exercise has a beneficial effect on cognitive functions or reduces an age related decline in these. Research on rodents suggest that an increase in memory and learning in relation to exercise is mediated through an up-regulation of brain derived neurotrophic factor, which has the ability to stimulate synaptic-plasticity.

Interestingly the exercise induced cell proliferation is inhibited by peripheral blockade of either insulin growth factor 1 (IGF-1) or vascular endothelial growth factor (VEGF), which could indicate that the exercise induced neurogenesis is dependent of IGF-I/VEGF. The role of IGF-I in neurogenesis is supported by studies showing an increase in new hippocampal cells in sedentary animals given IGF-I infusion. Fibroblast growth factor 2 (FGF-2) also increases in the rat hippocampus in response to exercise, however FGF-2 injections into the adult rat hippocampus do not increase neurogenesis. The importance of IGF-I in neurogenesis is emphasized by the fact that homozygous IGF1 -/- mice at the age of to months had reduced brain weight affecting all major brain areas, especially the volume of the dentate gyrus(33) in contrary to BDNF null mutant mice that did not show major hippocampal deficits.

Furthermore, it has been shown that antidepressant treatment up-regulates sBDNF in humans and a relationship between genetic variants of BDNF locus and depression have been implied. On this background it could be argued that low BDNF levels contribute to the pathophysiology of depression, and that exercise has a beneficial effect on cognitive function in patients with depression through an up-regulation of IGF-1, VEGF and BDNF.

The effect of exercise on hippocampal neurogenesis and cognition have recently been supported in a human study measuring cerebral blood volume in the dentate gyrus by magnetic resonance imaging.

On this background the investigators have designed this randomized trial comparing aerobic exercise and no treatment in light to moderate depression. This trial will employ adequate methods of reducing bias such as centralized randomization, blinded outcome assessment, and analysis according to the intent-to-treat principle. In addition the investigators plan to include a healthy control group to establish any differences in biological response to exercise

Objectives The primary objective for the DEMOII superiority trial is to assess the beneficial and harmful effect of aerobic exercise versus stretching exercise in patients diagnosed with moderate depression according to ICD-10. The primary outcome will be an assessment of depressive symptoms as measured with the Hamilton Depression Scale (HAM-D17), by outcome assessors blinded to intervention group.

The secondary objective is to measure the effect of exercise on neurogenesis in the hippocampal region by cerebral blood volume. The assessors will be blind to participation status.

Tertiary objects is to evaluate cognitive skills, brain derived neurotrophic factor, insulin like growth hormone 1, vascular endothelial growth factor, and other variables associated with the development of cardiovascular disease (interleukin 6, maximal oxygen uptake, BMI, tumour necroses factor alpha and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 60 years
2. Major depression according to DSM-IV
3. Living within 30 km of training facilities
4. Able to read and understand informed consent

Exclusion Criteria:

1. Recreational or current drug abuse
2. Having used antidepressant medication within the last 2 months
3. Contraindications to physical exercise
4. Recreational exercise> 1 hour per week
5. Medication for diabetes, hypertension, or any kidney disease
6. Suicidal behaviour (ham-d17 item3 > 2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
HAM-D17 | Before and after 3 months intervention

SECONDARY OUTCOMES:
Remission from depression (not fulfilling the DSM-IV criteria for depression and a hamilton rating below 8) | Before and after 3 months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Krogh, M.D, Principal Investigator — Psychiatric Center Bispebjerg, Bispebjerg University Hospital, Copenhagen Denmark
Locations (1):
- Psychiatric Center Bispebjerg, Copenhagen, Denmark

REFERENCES:
- [Derived] Krogh J, Rostrup E, Thomsen C, Elfving B, Videbech P, Nordentoft M. The effect of exercise on hippocampal volume and neurotrophines in patients with major depression--a randomized clinical trial. J Affect Disord. 2014 Aug;165:24-30. doi: 10.1016/j.jad.2014.04.041. Epub 2014 Apr 23. PMID 24882173
- [Derived] Krogh J, Videbech P, Thomsen C, Gluud C, Nordentoft M. DEMO-II trial. Aerobic exercise versus stretching exercise in patients with major depression-a randomised clinical trial. PLoS One. 2012;7(10):e48316. doi: 10.1371/journal.pone.0048316. Epub 2012 Oct 31. PMID 23118981